CLINICAL TRIAL: NCT00322218
Title: Phase III,Open-label,Prospective,Two-armed,Multicenter Study Comparing Zevalin Regimen With no Further Treatment in Patients With Diffuse Large B-cell Lymphoma.
Brief Title: Study Comparing Zevalin Regimen With no Further Treatment in Patients With Diffuse Large B-cell Lymphoma.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to low recruitment rate that would have led to a long study duration.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 307940/106-20
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Lymphoma, Large Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zevalin (Experimental): Patients received Zevalin.
  Zevalin Therapeutic Regimen:
  Day 1: Initial administration of 250 mg/m^2 rituximab, followed immediately by administration of 185 MBq of [111In]-ibritumomab tiuxetan ,in centers where centers where biodistribution imaging or dosimetry had not been required, the first rituximab infusion was given alone.
  - Day 7-9: Rituximab 250 mg/m^2, followed immediately by [90Y]-ibritumomab tiuxetan 14.8 MBq/kg given as a slow intravenous push over 10 minutes.
  Two treatment days one week apart were followed by a 12-week safety period.
  Interventions: Drug: Zevalin
- Observational (No Intervention): Patients in this arm did not receive any reference therapy; they remained free of any anti-lymphoma therapy and were observed for relapse. This was non-interventional Stage consisting of a longterm follow-up period (until completion of a median observation period of 5 years).

INTERVENTIONS:
Drug: Zevalin — Zevalin study treatment regimen consisted of 2 rituximab i.v. infusions (Day 1 and Day 7-9) and one [90Y]-ibritumomab tiuxetan infusion in connection with the second rituximab infusion.
  The core treatment regimen in the Zevalin arm was:
  Day 1: Rituximab i.v. infusion 250 mg/m^2
  Day 7-to 9: Rituximab i.v. infusion 250 mg/m^2 immediately followed by [90Y]-ibritumomab tiuxetan 14.8 MBq/kg (0.4 mCi/kg) with a maximum dose of 1184 MBq (32 mCi),administered as slow intravenous push over 10 minutes.
  Other Names: Ibritumomab tiuxetan
  Arms: Zevalin

SUMMARY:
This study treats patients with diffuse large B-cell lymphoma whose disease is in complete remission due to previous treatment with Cyclophosphamide Doxorubicin hydrochloride Vincristine Prednisolone- Rituximab (CHOP-R). Half of the patients received Zevalin and the other half receive no further anti-cancer treatment. The two patient groups compared to determine if Zevalin given after CHOP-R therapy provides greater benefits than receiving no additional anti-cancer therapy after CHOP-R.

DETAILED DESCRIPTION:
The objectives of this study were to evaluate the efficacy and safety of the Zevalin study regimen compared with observation alone in patients with complete remission (CR or CRu) after first-line CHOP-R, the study was to include patients 60-years-of-age or older with histologically confirmed Ann Arbor stage II, III, or IV diffuse large B-cell lymphoma

End Points:

Primary endpoint: Overall survival (OS) Secondary endpoints: Disease-free survival (DFS), health-related quality of life (HRQL) as assessed by the patient using standard questionnaires .

Number of Patients :

A total of 400 patients (200 per arm) were planned to be enrolled.

- In fact, 68 randomized patients (full analysis set; FAS) were analysed; 34 patients per each arm. The per-protocol set (PPS; 65 patients) comprised 33 patients allocated to the Zevalin arm and 32 patients allocated to the observation control arm.

Study Treatment :

The combination regimen with rituximab was designed in 2 steps as follows:

* Day 1: Initial administration of 250 mg/m^2 rituximab, followed immediately by administration of 185 megabecquerel (MBq) (5 millicurie [mCi]) of [111In]-ibritumomab tiuxetan (the latter one only in centers where biodistribution imaging or dosimetry was compulsory according to local law). In centers where biodistribution imaging or dosimetry had not been required, the first rituximab infusion was given alone.
* Day 7-9: Rituximab 250 mg/m^2, followed immediately by [90Y]-ibritumomab tiuxetan 14.8 megabecquerel/kilograms (MBq/kg) (0.4 millicurie / kilogram [mCi/kg]) (maximum dose 1184 MBq) given as a slow intravenous (I.V.) push over 10 minutes. Two treatment days one week apart followed by a 12-week safety period.

Duration of Patient Participation:

Due to the sequential design, the total duration of this study was not fixed. Originally, the study was planned in a randomized, parallel-group, group sequential design.

Objective :

The primary objective of this study was an inferential comparison between the 2 randomized groups in terms of overall survival using a group sequential triangular test ,since the study was prematurely terminated the pre-planned group-sequential nature of the study design was not applicable statistical analyses. Actually, the prominent efficacy variables for the OS and DFS were analysed in the FAS (identical to the safety analysis set) and PPS using Kaplan Meier estimates by treatment group.

Study Design :

This study was designed as a prospective, multi-center, open label, randomized, two-armed, group-sequential Phase III study. The study was planned to consist of 2 stages: an interventional Stage 1 with Screening/Baseline, treatment, safety, and follow-up periods, and a non-interventional Stage 2 consisting of a long-term follow-up period (until completion of a median observation period of 5 years). This second stage of the study was to be started only if superiority of the Zevalin study regimen could be demonstrated in the preceding Stage 1.

Pharmacokinetics/Pharmacodynamic results: Not applicable

Extent of exposure:

All 34 patients randomized to the Zevalin arm were given 2 rituximab infusions(with a median dose of 425.0 mg at each of the 2 infusion time points).Three patients underwent radioimaging studies/dosimetry and therefore were administered [111In]-ibritumomab tiuxetan at Day 1. All but 1 patient received an infusion with [90Y]-ibritumomab tiuxetan following the second infusion of rituximab. The mean dose ranged from 765.9 -1197.0 MBq.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, Ann Arbor stage II, III, or IV Diffuse large B-cell lymphoma (DLBCL) according to the Revised European American Lymphoma(REAL)/World Health Organization (WHO) classification .
* Central pathology review confirming the DLBCL diagnosis and Cluster of differentiation 20 (CD20) positivity, and no evidence of DLBCL in bone marrow
* First-line treatment of DLBCL must have been 6 or 8 cycles of standard CHOP chemotherapy in combination with rituximab .
* Complete remission(CR) or unconfirmed complete remission(CRu) according to the International Workshop Response Criteria for Non Hodgkins Lymphoma (NHL) described by Cheson et al and modified for this study after first-line treatment with CHOP-R. Computerised Tomography (CT) scans of chest, abdomen, pelvis, and neck (if applicable) must have been performed within 6 weeks after the last dose of the last course of CHOP-R. Applicability of the neck CT means that the patient had involvement of the neck region by palpation / physical examination at first diagnosis (pre-CHOP-R).
* Central radiographic review of the CT scans from before and after first-line treatment with CHOP-R fulfilling the radiological requirements for CR/CRu
* Patients 60 years of age or older at time of randomization
* WHO performance status (PS) of 0 to 2 within 1 week of randomization
* Absolute neutrophil count greater than or equal to 1.5 x 10^9/L within 1 week of randomization
* Hemoglobin greater than or equal to 10 g/dL within 1 week of randomization
* Platelets greater than or equal to 150 x 10^9/L within 1 week of randomization
* Life expectancy of 3 months or longer
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* Presence of any other malignancy or history of prior malignancy except non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma
* Prior radioimmunotherapy, radiation therapy, or any other NHL therapy except first-line CHOP-R
* Presence of gastric, central nervous system or testicular lymphoma at first diagnosis
* Histological transformation of low-grade non-Hodgkin's lymphoma (NHL)
* Known seropositivity for hepatitis C virus or hepatitis B surface antigen
* Known history of Human Immunodeficiency virus (HIV) infection
* Abnormal liver function: total bilirubin > 1.5 x upper limit of normal (ULN) or Alanine Aminotransferase > 2.5 x ULN within 1 week of randomization
* Abnormal renal function: serum creatinine > 2.0 x ULN within 1 week of randomization
* Nonrecovery from the toxic effects of CHOP-R therapy
* Known hypersensitivity to murine or chimeric antibodies or proteins
* Granulocyte Colony Stimulating Factor (G-CSF) or Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) therapy within two weeks (or four weeks if pegylated) prior to screening laboratory sampling
* Concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes,congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Male and female patients of child-bearing potential unwilling to practice effective contraception during the study and unwilling or unable to continue contraception for 12 months after their last dose of study treatment
* Female patients who are pregnant or are currently breastfeeding
* Treatment with investigational drugs less than 4 weeks before the planned Day 1 or nonrecovery from the toxic effects of such therapy
* Surgery less than 4 weeks before the planned Day 1 or nonrecovery from the side effects of such surgery
* Concurrent systemic corticosteroid use for any reason except as premedication in case of known or suspected allergies to contrast media or as premedication for potential side effects of rituximab treatment
* Unwillingness or inability to comply with the protocol

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (34):
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research site, Bakersfield, California
  - Research Site, Berkeley, California
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, Duarte, California
  - Research site, Los Angeles, California
  - Research site, Newport Beach, California
  - Research Site, San Diego, California
  - Research site, Vallejo, California
  - Research site, Aurora, Colorado
  - Research site, Newark, Delaware
  - Research site, St. Petersburg, Florida
  - Research Site, Coeur d'Alene, Idaho
  - Research site, Chicago, Illinois
  - Research site, Joliet, Illinois
  - Research Site, Morris, Illinois
  - Research site, Overland Park, Kansas
  - Research Site, Shreveport, Louisiana
  - Research site, Baltimore, Maryland
  - Research site, Boston, Massachusetts
  - Research site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Louis Park, Minnesota
  - Research Site, Commack, New York
  - Research Site, East Setauket, New York
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Aberdeen, South Dakota
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
- Austria (2):
  - Research Site, Graz
  - Research Site, Innsbruck
- Belgium (3):
  - Research Site, Bruges
  - Research Site, Ghent
  - Research Site, Leuven
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Oulu
- France (7):
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Cedax, Lyon
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (6):
  - Research Site, Chemnitz
  - Research Site, Jena
  - Research Site, Karlsruhe
  - Research Site, Mainz
  - Research Site, Rostock
  - Research Site, Würzburg
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Szeged
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Italy (5):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Torino
- Poland (4):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
- Research Site, Singapore, Singapore
- South Korea (2):
  - Research Site, Yonsei, Seoul
  - Research Site, Seoul
- Spain (4):
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Seville
- Sweden (3):
  - Research Site, Malmo
  - Research Site, Uddevalla
  - Research Site, Umeå
- Switzerland (2):
  - Research Site, Bern
  - Research Site, Sankt Gallen
- Research Site, Bangkok, Thailand
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diffuse large B-cell lymphoma (DLBCL) Patients at the age of at least 60 years and in complete remission (CR or CRu) after 6 or 8 cycles of a first-line treatment with Cyclophosphamide Doxorubicin hydrochloride Vincristine Prednisolone- Rituximab (CHOP-R) were enrolled in the study.
Pre-assignment Details: Of the 151 screened patients 68 patients were assigned to treatment (Full analysis set, FAS). Three patients showed major protocol deviations and thus were excluded from the "per protocol set"(PPS). The PPS comprised 65 patients.
Groups:
- Zevalin: Zevalin Therapeutic Regimen: Day 1: 250 milligram per meter square (mg/m^2) Rituxan followed by 5 millicurie (mCi) 111In Zevalin. Day 7: 250 mg/m^2 Rituxan followed by 0.4 millicurie/kilogram (mCi/kg) Zevalin.
- Observation: Patients in this arm were diagnosed with diffuse large B-cell lymphoma and were in complete remission after first-line CHOP-R therapy. Patients in this arm did not receive any reference therapy; they remained free of any anti-lymphoma therapy and were observed for relapse.
Period: Overall Study
Arm/Group | Zevalin | Observation
Started | 34 | 34
Per-Protocol Set | 33 | 32
Completed | 31 | 28
Not Completed | 3 | 6
Not completed — Death | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Zevalin: Zevalin Therapeutic Regimen: Day 1: 250 mg/m^2 Rituxan followed by 5 mCi 111In Zevalin. Day 7: 250 mg/m^2 Rituxan followed by 0.4 mCi/kg Zevalin.
- Total: Total of all reporting groups
Arm/Group | Zevalin | Observation | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 31 | 28 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (4.6) | 68.8 (4.8) | 69.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The primary analysis was based on the full analysis set (FAS). Actually, the prominent efficacy variable OS was analysed in the FAS (identical to the safety analysis set) and Per Protocol Set using Kaplan Meier estimates by treatment group. "Overall survival" was defined as the median time interval (in months)from randomization to death from any cause.This time-to-event variable was censored at the date of the last known follow-up visit (provided that the patient was still alive at that time).
Time Frame: 5 years or until patient dies or lost to follow up
Population: This study was completed in 2008. We have exhausted all efforts and unfortunately, the data cannot be located in our records. Therefore, no data is available to report for this outcome measure.
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion of Participants With Disease Free Survival (DFS)
Description: DFS was analysed in the FAS (identical to the safety analysis set) and Per Protocol set using Kaplan Meier estimates by treatment group.Disease-free survival was defined as the median time interval (in months) from randomization to the date of relapse (as assessed by the investigator) or death from any cause. This time-to-event variable was also censored at the date of the last known follow-up visit (provided that the patient was still alive at that time).
Time Frame: 5 years or until patient disease progresses or lost to follow up
Measure: Number; unit: proportion of participants
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 34 | 34
proportion of participants | 0.7058 | 0.7957
Statistical Analysis 1: Comparison: Zevalin vs Observation; Test type: Superiority or Other; p = 0.8578, Stratified Log-Rank Test

3. Secondary Outcome: The Health-related Quality of Life (HRQL)
Description: HRQL questionnaire consists of 27 questions each scores ranging from 0 - 4. The minimum score was 0 which is termed as 'worst imaginable health state' and the maximum score for a patient was 100 which is termed as 'best imaginable health state'.
  The descriptive classification defines health status in terms of 5 dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each dimension is subdivided into 3 levels: no problem, some or moderate problems, unable or extreme problems.
Time Frame: Up to Month 36
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Zevalin | Observation
Number analyzed (Participants) | 34 | 34
scores on a scale | 84.2 (14.2) | 88.7 (12.6)

ADVERSE EVENTS:
Time Frame: Followed up until last anti-lymphoma treatment or 42 months whichever is longer.
Description: Only study drug-related AEs was collected until the end of Stage 1 in case of a relapse.Patients who relapsed before study treatment were to be followed up in the same way as patients in observation arm,if a patient randomized to the observation arm received treatment for a relapse, no further AE reporting was required.
Arm/Group | Zevalin | Observation
Serious Adverse Events (participants affected / at risk) | 2/34 | 1/34
Other Adverse Events (participants affected / at risk) | 5/34 | 1/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=34) | Observation (N=34)
cytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin (N=34) | Observation (N=34)
Infections and manifestations (Infections and infestations) | 5 (5) | 1 (6)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated after 68 patients had been randomized due to a low recruitment rate that would have led to an unacceptably long study duration.No safety concerns or lack of efficacy had led to the decision to cancel the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No